CLINICAL TRIAL: NCT05641688
Title: An Open-label, Non-randomized, Multi-center Pivotal Phase 3 Study to Evaluate the Efficacy and Safety of PET Imaging With [18F]PI-2620 for the Detection of Tau Deposition When Compared to Post-mortem Histopathology (ADvance)
Brief Title: [18F]PI-2620 Phase 3 Histopathological Study
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Life Molecular Imaging Ltd (Industry)
Responsible Party: Sponsor
Organization: Life Molecular Imaging SA (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LMT-01-01-22
Record Dates: First submitted 2022-11-17; First posted 2022-12-08 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — ((18)F)PI-2620

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PI-2620 PET Scan (Experimental)
  Interventions: Drug: [18F]PI-2620

INTERVENTIONS:
Drug: [18F]PI-2620 — The radioligand, [18F]PI-2620, will be injected intravenously at a dose of 185 MBq ± 20%

SUMMARY:
This study is an open-label, multi-center, non-randomized pivotal Phase 3 study to assess the efficacy and safety of PET imaging with [18F]PI-2620 for detection of tau deposition in subjects with Alzheimer's disease (AD) and controls during lifetime when compared to histopathology obtained after death and completion of brain autopsy.

ELIGIBILITY:
Inclusion Criteria:

Only subjects who meet all of the following criteria will be eligible for enrollment into the study:

1. Males and females aged 50 years and over
2. Have a projected life expectancy of ≤ 1 year as determined by the investigator (terminal medical condition including but not limited to end-stage dementia, end-stage congestive heart failure, end-stage chronic obstructive pulmonary disease (COPD), or end-stage cancer)
3. Written informed consent obtained from the subject and/or the subject's legally authorized representative (LAR), as applicable, to consent for study procedures and brain donation (consent consistent with the legal requirements of the State in which the subject dies)
4. Can tolerate study procedures including lying down in PET scanner. The investigator will carefully assess each subject and use medical judgment to determine whether the subject can tolerate the imaging procedure

Exclusion Criteria:

Subjects will be excluded from the enrollment if they:

1. Are receiving aggressive treatment with life sustaining measures (e.g. receiving chemotherapy; palliative chemotherapy is allowed)
2. Are known to have a structural brain lesion that would interfere either with PET imaging or pathological assessment (e.g. lesions are typically > 2 cm at their greatest extent and may include stroke, primary or metastatic neoplasm, other tumors or cystic lesions. Subjects with a history of major stroke or traumatic brain injury or other structural lesion as well as cases with a history of primary Central Nervous System (CNS) neoplasm or known metastatic cancer must be discussed with the study sponsor prior to enrollment)
3. Have suspected encephalopathy due to alcoholism or end-stage liver disease
4. Are known to have a Glomerular Filtration Rate below < 15 mL/min
5. Have received an investigational or approved therapy directly targeting amyloid or tau
6. Are females of childbearing potential who are pregnant, lactating or breastfeeding, or who are not using adequate contraception
7. Have implants such as implanted cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, CNS aneurysm clips and other medical implants that have not been certified for MRI, or history of claustrophobia in MRI (in case an MRI is planned to be performed)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Efficacy of the visual assessment of [18F]PI-2620 PET imaging, in correctly differentiating tau neurofibrillary pathology associated with AD (NFT Score of B0 or B1 = negative) | At autopsy, until study completion with an average of 1 year
  [18F]PI-2620 PET scans will be classified as either tau-positive or tau-negative as defined by the reading methodology by each of the 5 independent readers blinded to the clinical and pathology information. NFT scores (as defined in Hyman et al. 2012) will be used as pathology assessment SoT (standard of truth). Tau neurofibrillary pathology associated with AD is defined as either negative with NFT Scores of B0 or B1 or positive NFT Scores of B2 or B3. The [18F]PI-2620 PET visual assessment will be compared with the pathology assessment to derive sensitivity and specificity estimates for each individual reader. Sensitivity and specificity are percentages that can range from 0 to 100%. The primary endpoint is considered to be met if for the same 3 out of 5 readers, the lower bound of the 95% CIs for both sensitivity and specificity are ≥ 50%.

SECONDARY OUTCOMES:
Diagnostic Efficacy of the visual assessment of [18F]PI-2620 PET imaging, in correctly differentiating tau neurofibrillary pathology associated with AD (NFT Score of B0, B1 or B2 = negative) | At autopsy, until study completion with an average of 1 year
  [18F]PI-2620 PET scans will be classified as either tau-positive or tau-negative as defined by the reading methodology by each of the 5 independent readers blinded to the clinical and pathology information. NFT scores (as defined in Hyman et al. 2012) will be used as pathology assessment SoT (standard of truth). Tau neurofibrillary pathology associated with AD is defined as either negative with NFT Scores of B0, B1 or B2 or positive NFT Scores of B3. The [18F]PI-2620 PET visual assessment will be compared with the pathology assessment to derive sensitivity and specificity estimates for each individual reader. Sensitivity and specificity are percentages that can range from 0 to 100%. The primary endpoint is considered to be met if for the same 3 out of 5 readers, the lower bound of the 95% CIs for both sensitivity and specificity are ≥ 50%.
Diagnostic efficacy of the visual assessment of [18F]PI-2620 PET imaging, in correctly differentiating levels of AD neuropathologic change (ADNC) ('No' or 'Low' levels of ADNC = negative) | At autopsy, until study completion with an average of 1 year
  [18F]PI-2620 PET scans will be classified as either tau-positive or tau-negative as defined by the reading methodology by each of the 5 independent readers blinded to the clinical and pathology information. ADNC levels according to NIA-AA criteria (Hyman et al., 2012) will be used as pathology assessment SoT (standard of truth). Level of ADNC according to NIA-AA criteria (considering Braak stage, Thal plaque score, and CERAD amyloid neuritic plaque score) is defined as either negative with 'no' or 'low' ADNC levels or positive with 'intermediate' or 'high' ADNC levels. The [18F]PI-2620 PET visual assessment will be compared with the pathology assessment to derive sensitivity and specificity estimates for each individual reader. Sensitivity and specificity are percentages that can range from 0 to 100%. The primary endpoint is considered to be met if for the same 3 out of 5 readers, the lower bound of the 95% CIs for both sensitivity and specificity are ≥ 50%.
Diagnostic efficacy of the visual assessment of [18F]PI-2620 PET imaging, in correctly differentiating levels of ADNC ('No', 'Low' or 'Intermediate" levels of ADNC = negative) | At autopsy, until study completion with an average of 1 year
  [18F]PI-2620 PET scans will be classified as either tau-positive or tau-negative as defined by the reading methodology by each of the 5 independent readers blinded to the clinical and pathology information. ADNC levels according to NIA-AA criteria (Hyman et al., 2012) will be used as pathology assessment SoT (standard of truth). Level of ADNC according to NIA-AA criteria (considering Braak stage, Thal plaque score, and CERAD amyloid neuritic plaque score) is defined as either negative with 'no', 'low' or 'intermediate' ADNC levels or positive with 'high' ADNC levels. The [18F]PI-2620 PET visual assessment will be compared with the pathology assessment to derive sensitivity and specificity estimates for each individual reader. Sensitivity and specificity are percentages that can range from 0 to 100%. The primary endpoint is considered to be met if for the same 3 out of 5 readers, the lower bound of the 95% CIs for both sensitivity and specificity are ≥ 50%.
Inter-reader agreement for the visual assessment of [18F]PI-2620 PET images | Baseline scan
  Fleiss kappa will be used to measure the inter-reader agreement for the visual assessment of [18F]PI-2620 PET images.

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Atri, MD, PhD, Principal Investigator — Banner Health; Andrew Stephens, MD, PhD, Study Director — Life Molecular Imaging
Locations (25):
- United States (25):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - UC Los Angeles, Los Angeles, California
  - Esperanza Clinical, Murrieta, California
  - Sutter Health, San Francisco, California
  - Galiz Research, Hialeah, Florida
  - UF College of Medicine - Jacksonville, Jacksonville, Florida
  - K2 Medical Research, Lady Lake, Florida
  - K2 Medical Research, Maitland, Florida
  - ClinCloud Research, Melbourne, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - The Roskamp Institute, Sarasota, Florida
  - Charter Research, Winter Park, Florida
  - Alzheimer's Disease Center, Braintree, Massachusetts
  - Headlands Research, Plymouth, Massachusetts
  - Be Well Clinical Studies, Lincoln, Nebraska
  - Darthmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Velocity Clinical Research, East Syracuse, New York
  - Ichor Research, Syracuse, New York
  - American Carolina Clinical Research LLC, Charlotte, North Carolina
  - Insight Clinical Trials LLC, Beachwood, Ohio
  - Valley Medical Research, Centerville, Ohio
  - Baylor Research Institute, Dallas, Texas
  - Sante Clinical Research, Kerrville, Texas
  - Be Well Clinical Studies, Round Rock, Texas

IPD SHARING:
Plan to Share IPD: Undecided